CLINICAL TRIAL: NCT04522453
Title: E-MhGAP Intervention Guide in Low- and Middle-income Countries: Proof-of-concept for Impact and Acceptability
Acronym: EMILIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Collaborators: King's College London (Other); Duke University (Other); Transcultural Psychosocial Organization Nepal (Other); University of Ibadan (Other); World Health Organization (Other); Medical Research Council (Other Government)
Responsible Party: Principal Investigator, Brandon A Kohrt, MD, PhD, Associate Professor, George Washington University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: MR/R023697/1
Record Dates: First submitted 2020-07-29; First posted 2020-08-21 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Depression
Keywords: Primary care; Competence; Mobile health; Mental health; Low- and middle-income countries; Training; Supervision
MeSH Terms: conditions — Depression; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Feasibility cluster randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Assessors will not be informed whether primary care providers or patients are in the paper of digital arm of the mental health Gap Action Program.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- paper mental health Gap Action Program-Intervention Guide (Active Comparator): This arm will be training and supervision as usual employing the standard paper version of the mental health Gap Action Program-Intervention Guide. Primary care workers will be trained to use the paper version of this tool and will use the paper version when evaluating patients.
  Interventions: Other: paper-based version of mental health Gap Action Program-Intervention Guide
- digital mental health Gap Action Program-Intervention Guide (Experimental): This arm will be training and supervision in an experimental approach using a digital version of version of the mental health Gap Action Program-Intervention Guide. The digital version allows for interactive decision making on diagnoses and care, and it allows for entering of patient data. Primary care workers in this arm will be trained to use the digital version of this tool and will use the digital version when evaluating patients.
  Interventions: Other: digital version of the mental health Gap Action Program-Intervention Guide

INTERVENTIONS:
Other: paper-based version of mental health Gap Action Program-Intervention Guide — A paper-based guide for diagnosis and management of mental disorders in primary care.
  Arms: paper mental health Gap Action Program-Intervention Guide
Other: digital version of the mental health Gap Action Program-Intervention Guide — A digital guide and client data entry tool for diagnosis and management of mental disorders in primary care.
  Arms: digital mental health Gap Action Program-Intervention Guide

SUMMARY:
Two strategies will be compared for training and supervising primary care workers delivering mental health services. Both strategies will use the World Health Organization mental health Gap Action Program-Intervention Guide. In the standard strategy, the paper-based version of the mental health Gap Action Program-Intervention Guide will be used. In the novel strategy an electronic version of the mental health Gap Action Program-Intervention Guide that can be used on mobile digital devices will be given to primary care workers. This is a feasibility cluster-randomized controlled trial to establish parameters for conducting a fully-powered cluster-randomized controlled trial comparing the paper versus digital strategy. The primary outcome of the subsequent fully powered trial will be the difference in accurate detection of depression.

DETAILED DESCRIPTION:
Mental illnesses are common, affecting one in every three people during their lifetimes. Globally, mental illnesses are the leading contributor of years lived with a disability. Despite the prevalence and impact of mental illness, a large difference between true and treated prevalence rates of mental disorders, also known as the mental health treatment gap, exists. It is estimated that more than 80% of people with severe mental illness in low and middle-income countries receive no treatment. Only 16.5% of people with depression living in low- and middle-income countries have access to minimally adequate treatment. The consequences of this treatment gap include symptom persistence and deterioration, social exclusion, and long-term disability of people who could be economically productive and socially included. Globally, there is growing recognition of the importance of mental health as evidenced by its inclusion in the 2030 United Nations Agenda for Sustainable Development and extension of the World Health Organization Comprehensive Mental Health Action Plan to 2030 by the World Health Assembly.

Limited numbers of mental health specialists and the concentration of care in hospital settings limits the availability and accessibility of care. Low treatment rates in low- and middle-income countries are related to poor demand and supply-side forces. High levels of stigma associated with mental illness manifest in low rates of help-seeking among those who would benefit from care. The World Health Organization recommends a task-shifting approach to strengthen the generalist workforce and improve access to health care, including mental health care. However, this requires the availability of evidence-based tools and appropriate training, supervision, and support.

In recent years there has been an exponential rise in global access to mobile technologies in low- and middle-income countries. In 2012 there were 287 million unique mobile phone subscribers across sub-Saharan Africa covering 32% of the population. Six years later, that number rose to 465 million representing 44% of the population. In Nepal, the number of mobile contracts surpasses the total population (26.49 million). The increased application of mobile technology to healthcare arena, known as mobile health (mobile-health), aims to provide a powerful platform to improve the quality of interventions employing a task-shifting approach and reduce the treatment gap. Mobile health (mobile-health) refers to the use of mobile technology in health interventions and service provision. In a recent World Health Organization survey, 87% of responding countries reported at least one government sponsored mobile-health programme in their country. However, only 14% of countries reported an evaluation of these programmes, raising concerns about insufficient evidence of impact.

A systematic review of smartphone use in clinical decision making by healthcare professionals identified seven randomised control trials conducted in high-income settings, which demonstrated improved knowledge, diagnosis, treatment decisions and documentation using mobile-health technology. Studies on mobile-health tools in low- and middle-income countries have had more mixed results. Improved compliance to protocols has been demonstrated with a smart phone tool in India. Conversely, a study in Uganda failed to show improvement in service user outcomes when community-based peer workers used mobile phones to communicate with supervisors. Qualitative data does, however, suggest the intervention facilitated task shifting and improved health worker morale.

In 2010, the World Health Organization launched the Mental Health Gap Action Programme Intervention Guide, an evidence-based assessment and management guide for mental, neurological and substance use conditions designed for use by primary and community health staff in low- and middle-income countries. The first edition of the mental health Gap Action Program-Intervention Guide has been implemented in over 100 countries. An updated version was launched in 2016 with new sections and updated evidence-based guidance. The mental health Gap Action Program-Intervention Guide v2.0 consists of eight modules addressing priority conditions (i.e. depression, psychoses, epilepsy, child and adolescent mental and behavioural disorders, dementia, disorders due to substance use, self-harm/suicide and conditions related to extreme stress). The guide provides an overview of common presentations for each condition followed by detailed guidance for assessment, management (including referral to specialist care) and follow-up.

The E-mental health Gap Action Program Intervention guide in Low and middle-income countries: proof-of-concept for Impact and Acceptability (Emilia) project seeks to re-address the treatment gap by developing a potentially practicable way for primary health care staff to monitor and treat people with mental illness according to evidence-based guidelines. The project is comprised of three phases: (1) development of an adapted e-mental health Gap Action Program intervention guide, (2) feasibility testing, and (3) knowledge transfer and future work.

Objectives

Emilia aims to test the feasibility of an electronic version of the mental health Gap Action Program-Intervention Guide v2.0 and trial procedures for the future evaluation of a large-scale trial, which would evaluate differences in depression detection between facilities using e-mental health Gap Action Program vs. paper mental health Gap Action Program. The objectives of this feasibility study, in preparation for a future trial, include the following:

1. To evaluate the feasibility and acceptability of primary care mental health services utilizing the e-mental health Gap Action Program-Intervention Guide for training, supervision, and delivery of care [primary objective];
2. To determine recruitment and retention rates for primary care workers and patients;
3. To establish the acceptability and feasibility of assessing primary health worker and patient outcomes;
4. To assess ethics and safety procedures using adverse event reporting;
5. To describe depression detection rates in primary health clinics; and
6. To describe depression treatment outcomes in primary health clinics.

ELIGIBILITY:
Inclusion Criteria:

* Primary Care Health Workers: Primary healthcare staff will be eligible to participate if they are employed by the primary care clinic or government and have roles and responsibilities that relate to the use of the mental health Gap Action Program (e.g. direct clinical use or supervision). All relevant primary care staff, regardless of individual study participation, will receive training in the mental health Gap Action Program. (electronic or paper version) and have ongoing remote support and supervision.
* Patients: Attending primary care for treatment; fluent in Nepali (for Nepal site) or Yoruba (for Nigeria site);

Exclusion Criteria:

* Primary Care Health Workers: No exclusion criteria.
* Patients: Adult attendees will be deemed ineligible for the study if they are unable to understand or complete study assessment (e.g. individuals with severe learning disability or dementia), unable give informed consent, or have a medical emergency requiring immediate intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3351 (Actual)
Dates: Start 2020-12-27 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Mental Health Gap Action Programme Depression Diagnosis Tool | Three months post training
  Unnabbreviated name of scale: "Mental Health Gap Action Programme Depression Diagnosis Tool"; Primary care health workers diagnosis of depression documented in clinical records; Unit of measure: % of patients with Mental Health Gap Action Programme Depression Diagnosis compared to number of patients with positive Patient Health Questionnaire depression screen

SECONDARY OUTCOMES:
Mental Health Gap Action Programme Depression Diagnosis Tool | One month prior to training
  Unnabbreviated name of scale: "Mental Health Gap Action Programme Depression Diagnosis Tool"; Primary care health workers diagnosis of depression documented in clinical records; Unit of measure: % of patients with Mental Health Gap Action Programme Depression Diagnosis compared to number of patients with positive Patient Health Questionnaire depression screen
Patient health questionnaire 9 | One month prior to training
  Unabbreviated scale title "Patient health questionnaire 9"; Self reported symptoms of depression; minimum 0, maximum 27; high score is worse outcome
Patient health questionnaire 9 | Three months post training
  Unabbreviated scale title "Patient health questionnaire 9"; Self reported symptoms of depression; minimum 0, maximum 27; high score is worse outcome
Patient health questionnaire 9 | Six months post training
  Unabbreviated scale title "Patient health questionnaire 9"; Self reported symptoms of depression; minimum 0, maximum 27; high score is worse outcome
World Health Organization Disability Assessment Schedule | One month pre training
  Unabbreviated name of scale: "World Health Organization Disability Assessment Schedule"; Self reported measure of functional impairment; Minimum score 0, Maximum 60; higher score is worse outcome
World Health Organization Disability Assessment Schedule | Three months post training
  Unabbreviated name of scale: "World Health Organization Disability Assessment Schedule"; Self reported measure of functional impairment; Minimum score 0, Maximum 60; higher score is worse outcome
World Health Organization Disability Assessment Schedule | Six months post training
  Unabbreviated name of scale: "World Health Organization Disability Assessment Schedule"; Self reported measure of functional impairment; Minimum score 0, Maximum 60; higher score is worse outcome
Mental health gap action program knowledge assessment | One day pre training
  Unabbreviated scale title: "Mental health gap action program knowledge assessment"; Multiple choice test of mental disorder diagnosis and management; Minimum score 0%, Maximum 100%, higher score is better outcome
Mental health gap action program knowledge assessment | One day post training
  Unabbreviated scale title: "Mental health gap action program knowledge assessment"; Multiple choice test of mental disorder diagnosis and management; Minimum score 0%, Maximum 100%, higher score is better outcome
Mental health gap action program knowledge assessment | Three months post training
  Unabbreviated scale title: "Mental health gap action program knowledge assessment"; Multiple choice test of mental disorder diagnosis and management; Minimum score 0%, Maximum 100%, higher score is better outcome
Mental health gap action program knowledge assessment | Eight months post training
  Unabbreviated scale title: "Mental health gap action program knowledge assessment"; Multiple choice test of mental disorder diagnosis and management; Minimum score 0%, Maximum 100%, higher score is better outcome
Enhancing Assessment of Common Therapeutic Factors | One day pre training
  Unabbreviated title: "Enhancing Assessment of Common Therapeutic Factors"; Objective structured clinical examination of common factors and diagnostic practices; Minimum=15, Maximum=60; higher score is better outcome
Enhancing Assessment of Common Therapeutic Factors | One day post training
  Unabbreviated title: "Enhancing Assessment of Common Therapeutic Factors"; Objective structured clinical examination of common factors and diagnostic practices; Minimum=15, Maximum=60; higher score is better outcome
Enhancing Assessment of Common Therapeutic Factors | Three months post training
  Unabbreviated title: "Enhancing Assessment of Common Therapeutic Factors"; Objective structured clinical examination of common factors and diagnostic practices; Minimum=15, Maximum=60; higher score is better outcome
Enhancing Assessment of Common Therapeutic Factors | Eight months post training
  Unabbreviated title: "Enhancing Assessment of Common Therapeutic Factors"; Objective structured clinical examination of common factors and diagnostic practices; Minimum=15, Maximum=60; higher score is better outcome
Social Distance Scale | One day pre training
  Unabbreviated scale title: "Social Distance Scale"; Self reported measure of stigma against persons with mental illness; Minimum score=12, Maximum Score=72; higher score is worse outcome
Social Distance Scale | One day post training
  Unabbreviated scale title: "Social Distance Scale"; Self reported measure of stigma against persons with mental illness; Minimum score=12, Maximum Score=72; higher score is worse outcome
Social Distance Scale | Three months post training
  Unabbreviated scale title: "Social Distance Scale"; Self reported measure of stigma against persons with mental illness; Minimum score=12, Maximum Score=72; higher score is worse outcome
Social Distance Scale | Eight months post training
  Unabbreviated scale title: "Social Distance Scale"; Self reported measure of stigma against persons with mental illness; Minimum score=12, Maximum Score=72; higher score is worse outcome
Enhancing Assessment of Common Therapeutic Factors - patient version | One month pre training
  Unabbreviated scale title: "Enhancing Assessment of Common Therapeutic Factors - patient version"; Patient report of primary care workers common factors skills; minimum score=0, maximum score=15; higher score is better outcome
Enhancing Assessment of Common Therapeutic Factors - patient version | Three months post training
  Unabbreviated scale title: "Enhancing Assessment of Common Therapeutic Factors - patient version"; Patient report of primary care workers common factors skills; minimum score=0, maximum score=15; higher score is better outcome
Enhancing Assessment of Common Therapeutic Factors - patient version | Six months post training
  Unabbreviated scale title: "Enhancing Assessment of Common Therapeutic Factors - patient version"; Patient report of primary care workers common factors skills; minimum score=0, maximum score=15; higher score is better outcome
Acceptability of Intervention Measure | Three months post training
  Unabbreviated scale title "Acceptability of Intervention Measure"; Subjective report of acceptability of intervention; A 5-item scale that measures the perception among implementation stakeholders that a given treatment, service, practice, or innovation is agreeable, palatable, or satisfactory. Minimum=5, Maximum=25; higher score is better
Acceptability of Intervention Measure | Eight months post training
  Unabbreviated scale title "Acceptability of Intervention Measure"; Subjective report of acceptability of intervention; A 5-item scale that measures the perception among implementation stakeholders that a given treatment, service, practice, or innovation is agreeable, palatable, or satisfactory. Minimum=5, Maximum=25; higher score is better
Acceptability of Intervention Measure - patient version | Six months post training
  Unabbreviated scale title "Acceptability of Intervention Measure"; Subjective report of acceptability of intervention; A 5-item scale that measures the perception among implementation stakeholders that a given treatment, service, practice, or innovation is agreeable, palatable, or satisfactory. Minimum=5, Maximum=25; higher score is better
Feasibility of Intervention Measure | Three months post training
  Unabbreviated title: " Feasibility of Intervention Measure"; Subjective report of feasibility of intervention; measures the extent to which a new treatment, or an innovation, can be successfully used or carried out within a given agency or setting. Minimum=5, Maximum=25; higher score is better
Feasibility of Intervention Measure | Eight months post training
  Unabbreviated title: " Feasibility of Intervention Measure"; Subjective report of feasibility of intervention; measures the extent to which a new treatment, or an innovation, can be successfully used or carried out within a given agency or setting. Minimum=5, Maximum=25; higher score is better
Intervention Appropriateness Measure | Three months post training
  Unabbreviated title: " Intervention Appropriateness Measure"; Subjective report of appropriateness of intervention; A 5-item scale that measures the perceived fit, relevance, or compatibility of the innovation or evidence-based practice for a given practice setting, provider, or consumer, and/or perceived fit of the innovation to address a particular issue or problem. Minimum=5, Maximum=25; higher score is better
Intervention Appropriateness Measure | Eight months post training
  Unabbreviated title: " Intervention Appropriateness Measure"; Subjective report of appropriateness of intervention; A 5-item scale that measures the perceived fit, relevance, or compatibility of the innovation or evidence-based practice for a given practice setting, provider, or consumer, and/or perceived fit of the innovation to address a particular issue or problem. Minimum=5, Maximum=25; higher score is better
Intervention Appropriateness Measure - patient version | Six months post training
  Unabbreviated title: " Intervention Appropriateness Measure"; Subjective report of appropriateness of intervention; A 5-item scale that measures the perceived fit, relevance, or compatibility of the innovation or evidence-based practice for a given practice setting, provider, or consumer, and/or perceived fit of the innovation to address a particular issue or problem. Minimum=5, Maximum=25; higher score is better
Organizational Readiness for Implementing Change | One day pre training
  Unabbreviated title: "Organizational Readiness for Implementing Change"; Subjective report of readiness for implementing a new intervention; a 16-item tool to assess Assesses perspectives on intra- and extra-organizational implementation readiness; minimum=16, maximum=90; higher score is better
Normalization Measure Development | Eight months post-training
  Unabbreviated title: "Normalization Measure Development"; Subjective report of normalization of measure development; a brief self-report questionnaire that could be helpful in measuring implementation progress. Based on the Normalization Process Theory, this instrument focuses on 4 generative mechanisms involved in implementation processes: coherence, cognitive participation, collective action, and reflexive monitoring. 20 items; minimum=20, maximum=100, higher score is better outcome
Perceptions of supervisory support scale | Eight months post-training
  Unabbreviated title: "Perceptions of supervisory support scale"; Health workers perception of supervision support; 19 items, minimum score=19, maximum score=95; higher score is better outcome
Depression Attitudes Questionnaire | One day pre training
  Unabbreviated title:"Depression Attitudes Questionnaire"; Health workers report of attitudes toward depression care; Minimum=10; Maximum=40, higher scores=better outcome
Depression Attitudes Questionnaire | One day post training
  Unabbreviated title:"Depression Attitudes Questionnaire"; Health workers report of attitudes toward depression care; Minimum=10; Maximum=40, higher scores=better outcome
Depression Attitudes Questionnaire | One month post training
  Unabbreviated title:"Depression Attitudes Questionnaire"; Health workers report of attitudes toward depression care; Minimum=10; Maximum=40, higher scores=better outcome
Depression Attitudes Questionnaire | Three months post training
  Unabbreviated title:"Depression Attitudes Questionnaire"; Health workers report of attitudes toward depression care; Minimum=10; Maximum=40, higher scores=better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Graham Thornicroft, MD, PhD, Principal Investigator — King's College London
Locations (2):
- Transcultural Psychosocial Organization Nepal, Kathmandu, Nepal
- University of Ibadan, Ibadan, Oyo State, Nigeria

IPD SHARING:
Plan to Share IPD: Yes
An individual participant data sharing plan will address both primary care health worker and patient data.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: An individual participant data sharing plan and approach will developed for sharing after dissemination of the primary findings.
Access Criteria: Contact study investigators with data request.

REFERENCES:
- [Derived] Kohrt BA, Ojagbemi A, Luitel NP, Bakolis I, Bello T, McCrone P, Taylor Salisbury T, Jordans MJD, Votruba N, Carswell K, Green E, Gkaintatzi E, Lamichhane B, Elugbadebo O, Kola L, Lempp H, Chowdhary N, Dua T, Gureje O, Thornicroft G. An App-Based WHO Mental Health Guide for Depression Detection: A Cluster Randomized Clinical Trial. JAMA Netw Open. 2025 May 1;8(5):e2512064. doi: 10.1001/jamanetworkopen.2025.12064. PMID 40408108
- [Derived] Taylor Salisbury T, Kohrt BA, Bakolis I, Jordans MJ, Hull L, Luitel NP, McCrone P, Sevdalis N, Pokhrel P, Carswell K, Ojagbemi A, Green EP, Chowdhary N, Kola L, Lempp H, Dua T, Milenova M, Gureje O, Thornicroft G. Adaptation of the World Health Organization Electronic Mental Health Gap Action Programme Intervention Guide App for Mobile Devices in Nepal and Nigeria: Protocol for a Feasibility Cluster Randomized Controlled Trial. JMIR Res Protoc. 2021 Jun 15;10(6):e24115. doi: 10.2196/24115. PMID 34128819